CLINICAL TRIAL: NCT06720155
Title: The Effects of a Sleeper Stretch Intervention on Measures of Performance and Pain in CrossFit Participants: A Randomized Trial
Brief Title: Sleeper Stretch in CrossFit Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alecia M. Gende, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-007771
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Shoulder Pain
Keywords: CrossFit; Sleeper stretch
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleeper Stretch (Experimental)
  Interventions: Behavioral: Sleeper stretch
- Control Group (Active Comparator)
  Interventions: Behavioral: Standard workout

INTERVENTIONS:
Behavioral: Sleeper stretch — Participants will complete their regularly scheduled workout activities over 8 weeks, with the addition of the sleeper stretch into the dynamic warm-up. Participants will be instructed to lie side-lying with the dominant arm downward, the trunk rotated posteriorly 20 to 30°, the shoulder raised to 90°, the elbow flexed to 90°, and both knees semi-flexed to ensure stability. Participants will then be asked to use the opposite hand to grasp the dominant hand below the wrist and gradually internally rotate the forearm towards the floor; (i.e., the participant will perform passive internal rotation with the opposite arm). This stretch position will be completed on both sides. Participants will be instructed to complete 2 sets of 10 repetitions for each arm and hold the position for ~2 seconds.
  Arms: Sleeper Stretch
Behavioral: Standard workout — Participants will complete their regularly programmed dynamic warm-ups before scheduled workout for 8 weeks.
  Arms: Control Group

SUMMARY:
The purpose of this study is to compare the efficacy of the sleeper stretch in improving shoulder range of motion, strength and upper body performance in CrossFit athletes.

ELIGIBILITY:
Inclusion Criteria:

• Regularly active (attending CrossFit > 2x per week)

Exclusion Criteria:

* Positive test for labral lesions or rotator cuff tears
* History of recent fracture
* Orthopedic surgery in the upper limbs or cervical region
* Any other current injury that would prevent participation in regular work-shift activities

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Upper body function | Baseline, 4 weeks, 8 weeks
  Measured by isometric horizontal push test (IHPT), a newly designed test that selectively measures the horizontal component of maximal isometric force, with 3 minutes of rest between each trial. The participants will place their hands on force platforms that sample ground reaction force data at 1000 Hz throughout the test.

CONTACTS AND LOCATIONS:
Overall Officials: Alecia Gende, DO, CAQSM, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Health System-La Crosse, La Crosse, Wisconsin
  - Driftless CrossFit, Onalaska, Wisconsin

IPD SHARING:
Plan to Share IPD: No